CLINICAL TRIAL: NCT04486196
Title: Effect of Root Canal Disinfection With 980 µm Diode Laser on Post-operative Pain After Endodontic Treatment in Teeth With Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Effect of Diode Laser on Post-operative Pain After Endodontic Treatment in Teeth With Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Sema Sönmez Kaplan, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BİRUNİ-BAP-01-01
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Apical Periodontitis; Postoperative Pain
Keywords: diode laser; irrigation; post-operative pain; root canal treatment; visual analog scale
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative | interventions — Biodent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Laser) Group (Experimental): The final irrigation was performed using 5ml 2.5% NaOCI, followed by 5 ml 17% EDTA for 3 min and 5 ml distilled water.
  Interventions: Procedure: 2.5% NaOCl, %17 EDTA, Distilled water, 30-gauge, side-opening needle (Canal Clean, Biodent, South Korea),
- Laser Disinfection (LD) Group (Experimental): After final irrigation was performed using 5ml 2.5% NaOCI, followed by 5 ml 17% EDTA for 3 min and 5 ml distilled water, root canals were irradiated with 980 nm diode laser coupled with optical fiber 200 µm with setting at the average power 1.2-W in pulsed mode. 10 seconds irradiation followed by 10 seconds pause, which comprised one lasting cycle. This cycle was applied 4 times for each root canal. The optical fiber (Medency) was inserted 1 mm short of the apex and the root canals were slowly (at a speed of 2mm/s) irradiated from apical to coronal in continuous circling movements to treat all dentinal tubules in one cycle for each power.
  Interventions: Device: Medency Primo Diode Laser Device (Medency, Vicenza, Italy)

INTERVENTIONS:
Device: Medency Primo Diode Laser Device (Medency, Vicenza, Italy) — Root canals were irradiated with 980 nm diode laser coupled with optical fiber 200 µm with setting at the average power 1.2-W in pulsed mode. 10 seconds irradiation followed by 10 seconds pause, which comprised one lasting cycle.
  Arms: Laser Disinfection (LD) Group
Procedure: 2.5% NaOCl, %17 EDTA, Distilled water, 30-gauge, side-opening needle (Canal Clean, Biodent, South Korea), — Final conventional irrigation
  Arms: Control (No Laser) Group

SUMMARY:
Aim: This study aims to assess the effect of root canal disinfection with a 980 µm diode laser following chemomechanical root canal preparation on the severity of pain after root canal treatment (RCT).

Materials and Methods: In present study, asymptomatic, single-rooted teeth with periapical index (PAI) score 3 or 4 were included. All patients were treated with two visits of root canal treatment including dressing with calcium hydroxide. Patients were randomly divided into two groups (n: 28). 'Control (no laser)': The final irrigation was performed using 5ml 2.5% NaOCI, followed by 5 ml 17% EDTA and 5 ml distilled water. 'Laser Disinfection (LD)': Root canals were irradiated with 980 µm diode laser after final irrigation at both visits. The pain levels were evaluated using visual analog scale (VAS) after 8, 24, 48 hours and 7 days. In addition, analgesic intake and time intervals were recorded by patients. The collected data were statistically analyzed with the Chi-square and Mann-Whitney U test (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Patients that had asymptomatic, single-rooted teeth with PAI score 3 or 4

Exclusion Criteria:

* antibiotic use with in the last month,
* anti-inflammatory analgesic use within the last five days,
* systemic disorder, pregnancy or lactation,
* traumatic occlusion,
* presence of other teeth requiring RCT,
* teeth with root canal fillings,
* calcified canals,
* root resorption,
* periodontal diseases,
* sinus tracts
* severe crown destruction preventing rubber-dam application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-11-02 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 7 days
  Post-operative pain levels in each group will be assessed by visual analog scale (VAS).The pain levels will be evaluated after 8, 24, 48 hours and 7 days.

SECONDARY OUTCOMES:
Analgesic intake | 7 days
  After first and second appointments, analgesic use and time intervals will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Sönmez Kaplan, DDS, PhD, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not decided which collected IPD or which IPD that underlie results to share in a publication.

REFERENCES:
- [Derived] Kaplan T, Sezgin GP, Sonmez Kaplan S. Effect of a 980-nm diode laser on post-operative pain after endodontic treatment in teeth with apical periodontitis: a randomized clinical trial. BMC Oral Health. 2021 Jan 22;21(1):41. doi: 10.1186/s12903-021-01401-w. PMID 33482797